CLINICAL TRIAL: NCT00840242
Title: Smoking Reduction or Cessation With Nicotine Replacement Therapy. A Placebo Controlled Double Blind Trial With Nicotine Gum or Inhaler.
Brief Title: Smoking Reduction or Cessation With Nicotine Replacement Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: McNeil AB (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 97 NITG 001
Record Dates: First submitted 2009-02-09; First posted 2009-02-10 (Estimated); Last update posted 2012-04-25 (Estimated); Status verified 2012-04

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Nicotine Chewing Gum; Nicotine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Nicotine gum (Experimental): Nicotine gum
  Interventions: Drug: Nicotine gum
- Placebo gum (Placebo Comparator): Placebo gum
  Interventions: Drug: Placebo gum
- Nicotine inhaler (Active Comparator): Nicotine inhaler
  Interventions: Drug: Nicotine inhaler
- Placebo inhaler (Placebo Comparator): Placebo inhaler
  Interventions: Drug: Placebo inhaler

INTERVENTIONS:
Drug: Nicotine gum — 8-12 pieces per day, maximum 24 daily
  Other Names: Nicorette® Gum
  Arms: Nicotine gum
Drug: Placebo gum — 8-12 pieces per day, maximum 24 daily
  Arms: Placebo gum
Drug: Nicotine inhaler — 6-12 cartridges per day, maximum 12 daily
  Other Names: Nicorette® Inhaler
  Arms: Nicotine inhaler
Drug: Placebo inhaler — 6-12 cartridges per day, maximum 12 daily
  Arms: Placebo inhaler

SUMMARY:
The purpose of this study is to test the success rate of smoking reduction or cessation with different nicotine products.

DETAILED DESCRIPTION:
To test if smoking reduction or cessation is induced with different nicotine products and to investigate the possible health benefits of smoking reduction

ELIGIBILITY:
Inclusion Criteria:

* Age above 18
* Smoking >/= 15 cigarettes/day
* Having smoked for 3 years or more
* CO >/= 10ppm at inclusion
* Want to reduce smoking
* Prepared to adhere to the protocol
* Willing to provide signed informed consent
* Having made at least one serious attempt to quit smoking

Exclusion Criteria:

* Unstable angina pectoris, myocardial infarction within the last three months
* Use of other nicotine-containing products such as cigars, pipes, snuff
* Current use of NRT or involved in behavioral or pharmacological smoking cessation/reduction program
* Pregnancy/lactation or intended pregnancy
* Under psychiatric care or medication that might interfere with the trial
* Abuse of alcohol or any other drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 314 (Actual)
Dates: Start 1999-02; Primary Completion 2000-05 (Actual); Study Completion 2000-05 (Actual)

PRIMARY OUTCOMES:
Reduction in number of smoked cigarettes/day verified by carbon monoxide (CO) levels | Baseline to 6 weeks, 3 and 4 months

SECONDARY OUTCOMES:
Changes in laboratory values of cardiovascular risk factors | Baseline up to 12 months
Changes in clinical and laboratory exposure parameters | Baseline up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Kruse, PhD, Study Director — McNeil AB
Locations (2):
- Czechia (2):
  - Smoking Cessation Clinic, Kutná Hora
  - Institute of Hygiene and Epidemiology, Prague